CLINICAL TRIAL: NCT03454113
Title: Ellipsys Vascular Access System Registry, Protocol 1.0. Version 1.0
Brief Title: Ellipsys Vascular Access System Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 1.0 ver 1.0 23 January 2017
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-11

CONDITIONS: End-stage Renal Disease
Keywords: dialysis autogenous arterio-venous fistula
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Ellipsys Vascular Access — The Ellipsys Vascular Access System comprises the Ellipsys Catheter, Ellipsys Crossing Needle and Ellipsys Power Controller. The Ellipsys Crossing Needle is used to facilitate access between the artery and the vein. The Ellipsys Catheter is placed percutaneously into the selected vein in close proximity to the selected artery. The Ellipsys Catheter is actuated at the selected anastomosis site, and the vein and artery are approximated. Once the vessels are in the appropriate relative positions the catheter is connected to the Ellipsys Power Controller to create the anastomosis after which the Ellipsys Catheter is removed, and the access site is closed using standard percutaneous closure techniques.

SUMMARY:
Ellipsys Vascular Access System Registry will enroll up to 100 patients to evaluate the use and performance of the Ellipsys Vascular Access System when it is used within its intended use in accordance with standard of care in a clinical setting. The Ellipsys Vascular Access System is intended for use to create an arteriovenous (AV) fistula via percutaneous access.

DETAILED DESCRIPTION:
Ellipsys Vascular Access System Registry is a non-randomized, prospective, post-market, multi-center registry of the Ellipsys Vascular Access System in which up to 100 patients will be enrolled to evaluate the use and performance of the Ellipsys Vascular Access System when it is used within its intended use in accordance with standard of care in a clinical setting. The Ellipsys Vascular Access System is intended for use to create an AV fistula via percutaneous access. The primary performance endpoint is Clinical Success at the 90-day endpoint, where Clinical Success is defined as an access site that achieves a venous diameter of greater than or equal to 4 mm and blood flow greater than or equal to 500 ml/min in the brachial artery as measured via duplex ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with End-Stage Renal Disease (ESRD) or chronic kidney disease requiring dialysis or anticipated start of dialysis within 6 months of enrollment.
* Patients deemed medically eligible for upper extremity autogenous AV fistula creation, per institutional guidelines and/or clinical judgment Adequate quality vein base on pre-operative assessment:

  1. Vein diameter of > 2.0 mm at target anastomosis site
  2. Clinically significant outflow as determined by outflow mapping (ultrasound or v venography)
* Adequate quality artery base on pre-operative assessment:

  1. Arterial lumen diameter of > 2.0 mm at target anastomosis site
  2. No significant calcification at the anastomosis site
  3. Radial artery at the wrist suitable for catheterization
* Radial artery-adjacent vein proximity < 1.5 mm measured lumen edge-to-lumen edge as determined by pre-procedural ultrasound and confirmed pre-procedure
* Patent palmar arch with adequate collateral perfusion as evidenced by Negative Allen's Test
* Able and willing to follow a daily aspirin and/or other anticoagulation/antiplatelet regimen, not including warfarin (Coumadin, or comparable anti-coagulant)

Exclusion Criteria:

* Documented or suspected central venous stenosis including upper extremity arterial stenosis (≥ 50%)
* History of steal syndrome from a previous hemodialysis vascular access on the ipsilateral side which required intervention or abandonment
* Evidence of clinically significant vascular disease at the radial artery/adjacent vein site on the ipsilateral side
* Systolic pressures < 100 mg Hg at the time of treatment
* Suspected or confirmed skin disease at the skin entry site
* Immunocompromised patients (e.g. HIV positive)
* Edema of the upper extremity on the ipsilateral side
* Patients requiring immunosuppressant therapy such as Sirolimus (Rapamune®) or - Prednisone at a dose of > 10 mg per day
* Peripheral white blood cell count <1.5 K/mm3 or platelet count <75,000 cells/mm3
* Known bleeding diathesis or coagulation disorder
* Receiving warfarin (Coumadin, or comparable anti-coagulant) therapy
* Patients with acute or active infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with End-Stage Renal Disease or chronic kidney disease who provide written informed consent; who are currently require dialysis or it is anticipated will need dialysis within six months of enrollment; who meet all inclusion criteria and none of the exclusion criteria; and who are considered eligible for enrollment.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
The number of patients with a vascular access site that achieves a venous diameter of greater than or equal to 4 mm and blood flow greater than or equal to 500 ml/min in the brachial artery as measured via duplex ultrasound. | 90 days
  Primary endpoint

SECONDARY OUTCOMES:
Percent of Ellipsys Vascular Access procedures that successfully create an arteriovenous fistula (AVF) excluding Access Failures. | 12 months
  Device Success Rate
The length of time until a patient is able to undergo 2-needle cannulation for dialysis OR access vessel has a diameter ≥ 6 mm and a mean flow rate of ≥ 600 ml/min if the patient is not undergoing dialysis. | 12 months
  Time to Functional Patency
Percent of patients that require dialysis and sustain 3 consecutive 2-needle cannulations at the prescribed needle gauge and blood flow rate. | 12 months
  Dialysis Rate
The number of surgical or endovascular interventions required to achieve or maintain Functional Patency. | 12 months
  Secondary Procedure Rate
Number of patients with patency defined as an anastomosis that has flow whether it is being used for dialysis or not. | 12 months
  Arterio-venous fistula patency
Length of time from initial access creation to achieve Functional Patency or to time of abandonment of AVF. | 12 months
  Cumulative patency

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum des Saarlandes, Saarbrücken
  - Ammerland Klinik, Westerstede